CLINICAL TRIAL: NCT01810042
Title: A Prospective, Interventional Case Series, Effect of Lucentis on Indocyanine Angiographic Changes in Patients With Wet Age-related Macular Degeneration
Brief Title: Indocyanine Angiographic Changes of Choroidal Neovascularization by Ranibizumab
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Ji Eun Lee, Associate professor, Pusan National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 임상20120178
Record Dates: First submitted 2013-03-11; First posted 2013-03-13 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-03

CONDITIONS: Exudative Age-related Macular Degeneration
Keywords: age-related macular degeneration; choroidal neovascularization; ranibizumab; indocyanine angiography
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Ranibizumab; lactitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ranibizumab (Experimental): 0.5mg of ranibizumab is injected into the vitreous cavity monthly 3 times for the 3 months then pro-re-nata (PRN) for following 3 months.
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab — 0.5mg of ranibizumab is injected into the vitreous cavity through pars plana.
  Other Names: intravitreal injection of ranibizumab (Lucentis, Novartis)

SUMMARY:
Exudative age-related macular degeneration (ARMD) is complicated by choroidal neovascularization (CNV). Although anti-vascular endothelial growth factor treatment is the gold standard treatment, recurrence is the main limitation of the treatment. The changes of the CNV vascular structure is expected to provide information regarding recurrence. In the eyes that the vascular structure is clearly seen in indocyanine green angiography (ICGA), the vascular changes after ranibizumab injections will be investigated prospectively.

DETAILED DESCRIPTION:
For patients having exudative ARMD with CNV, whose vascular structures are clearly demonstrated in ICGA , ranibizumab is injected monthly three times, then pro re nata to 6 months. Vascular structures of CNV is investigated at baseline, 3 and 6 months using ICGA. Expected number of patients are 48 eyes from 4 centers, competitively.

ELIGIBILITY:
Inclusion Criteria:

1. age >= 50
2. Visual acuity of the study eye is between 20/400 and 20/40, and the other eye is 20/400 or better
3. Area of choroidal new vessel (CNV) clearly visible in indocyanine green angiography (ICGA) is more then 1/2 disc area.
4. Area of CNV clearly visible in ICGA is more than half of the total CNV area.

Exclusion Criteria:

1. CNV caused by other than age-related macular degeneration. (polypoidal choroidal vascularization, retinal angiomatous proliferation, degenerative myopia etc)
2. Blocked fluorescence in ICGA is more than half of the total CNV area.
3. Disciform scar
4. Previous anti-vascular endothelial growth factor (VEGF) treatment within 3 months
5. Previous any treatment of photodynamic therapy or photocoagulation
6. Previous intraocular or periocular injection of steroid within 3 months
7. Previous intraocular surgery except cataract surgery
8. Vitreo-retinal interface disease on the macula
9. Presence of other diseases may affect visual acuity (uveitis, glaucoma, diabetic retinopathy, etc.)
10. Uncontrolled periocular or intraocular infection
11. History of hypersensitivity to ranibizumab treatment
12. Uncontrolled systemic diseases (hypertension, diabetes mellitus, etc.)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ji Eun Lee, MH, PhD, Principal Investigator — Pusan National Universtiy Hospital
Locations (2):
- South Korea (2):
  - Pusan National University Hospital, Busan
  - Haeundae Baik Hospital, Busan

REFERENCES:
- [Background] Wong TY, Knudtson MD, Klein R, Klein BE, Meuer SM, Hubbard LD. Computer-assisted measurement of retinal vessel diameters in the Beaver Dam Eye Study: methodology, correlation between eyes, and effect of refractive errors. Ophthalmology. 2004 Jun;111(6):1183-90. doi: 10.1016/j.ophtha.2003.09.039. PMID 15177969
- [Background] Rosenfeld PJ, Brown DM, Heier JS, Boyer DS, Kaiser PK, Chung CY, Kim RY; MARINA Study Group. Ranibizumab for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1419-31. doi: 10.1056/NEJMoa054481. PMID 17021318
- [Background] Brown DM, Kaiser PK, Michels M, Soubrane G, Heier JS, Kim RY, Sy JP, Schneider S; ANCHOR Study Group. Ranibizumab versus verteporfin for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1432-44. doi: 10.1056/NEJMoa062655. PMID 17021319
- [Background] Spaide RF. Rationale for combination therapies for choroidal neovascularization. Am J Ophthalmol. 2006 Jan;141(1):149-56. doi: 10.1016/j.ajo.2005.07.025. PMID 16386991

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 53 patients were screened and 49 patients were enrolled from Oct 2010 to Feb 2013 in Pusan National University Hospital and Inje Baik Haeundae Hospital.
Pre-assignment Details: This study has a single arm, and there was no assignment process.
Groups:
- Ranibizumab: Ranibizumab is injected monthly 3 times then pro re nata (PRN) to 6 months.
  intravitreal injection of ranibizumab: 0.5mg of ranibizumab is injected into the vitreous cavity through pars plana.
Period: Overall Study
Arm/Group | Ranibizumab
Started | 49
Completed | 39
Not Completed | 10
Not completed — Lost to Follow-up | 10

BASELINE CHARACTERISTICS:
Population: Of 39 patients completed the study, 8 patients were excluded because 6 patients had polypoidal choroidal vasculopathy, and 2 patients had poor quality of indocyanine green angiography.
Groups:
- Ranibizumab: Ranibizumab is injected monthly 3 times then PRN to 6 months.
  intravitreal injection of ranibizumab: 0.5mg of ranibizumab is injected into the vitreous cavity through pars plana.
Arm/Group | Ranibizumab
Number analyzed (Participants) | 31
Age, Continuous [Mean (Full Range); unit: years] | 69 [51 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 19
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 31
Median visual acuity (ETDRS) [Median (Full Range); unit: ETDRS letter] — Visual acuity was measured using a Early Treatment of Diabetic Retinopathy Study (ETDRS) chart. The ETDRS score represents the number of letters that the patient read correctly. It can be ranged from 0 to 85. An ETDRS score of 85 corresponds to 20/20 vision approximately, and a score of 35 corresponds to 20/200 vision.
  ETDRS letter | 46 [0 to 81]
Central subfield macular thickness (um) [Median (Full Range); unit: micrometer] | 317 [168 to 793]

OUTCOME MEASURES:

1. Primary Outcome: Caliber of Choroidal New Vessel (CNV)
Description: Caliber of the largest CNV is measured using a software of IVAN (developed by Wisconsin University) that measures a caliber of retinal vessels using a semi-automatic method. An indocyanine green angiography (ICGA) image showing the vascular structures of CNV was processed to invert black and white for the analysis. The image was loaded in the software, and the course of the arteriolar CNV was indicated manually. Then average thickness of the vascular segment was calculated.
Time Frame: 6 months
Population: Of 31 patients included in the baseline analysis, 7 patients had the thickest vessels under limitation of measurement.
Measure: Mean (Full Range); unit: micrometer
Arm/Group | Ranibizumab
Number analyzed (Participants) | 24
micrometer | 43.53 [28.79 to 99.40]

2. Secondary Outcome: Lesion Size of CNV
Description: Lesion size of CNV is measured in fluorescein angiography using software, and find correlation with caliber of choroidal new vessels.
Time Frame: 6 months
Population: Among 39 patients who completed the study, 8 patients were excluded because of poor ICGA quality or presence of polypoidal choroidal vasculopathy.
Measure: Mean (Full Range); unit: square milimeter
Arm/Group | Ranibizumab
Number analyzed (Participants) | 31
square milimeter | 3.03 [0.07 to 18.09]

3. Secondary Outcome: Visual Acuity in ETDRS Letters
Description: Visual acuity was assessed using the ETDRS chart. The ETDRS chart includes 100 letters as the maximum possible score, and 0 letters read as the minimum possible score. Higher scores represents better functioning.
Time Frame: 6 months
Population: as for outcome 2
Measure: Median (Full Range); unit: ETDRS letters
Arm/Group | Ranibizumab
Number analyzed (Participants) | 31
ETDRS letters | 69 [2 to 90]

4. Secondary Outcome: Visual Acuity Changes
Description: Visual acuity is measured at baseline and 6 months using ETDRS chart. The changes was calculated by visual acuity at 6 months minus visual acuity at baseline.
  Positive values represent improvement of visual acuity, and negative values represent worsening of visual acuity at 6 months compared to baseline.
Time Frame: baseline and 6 months
Population: as for outcome 2
Measure: Median (Full Range); unit: ETDRS letters
Arm/Group | Ranibizumab
Number analyzed (Participants) | 31
ETDRS letters | 12.5 [-36 to 90]

ADVERSE EVENTS:
Arm/Group | Ranibizumab
Serious Adverse Events (participants affected / at risk) | 2/49
Other Adverse Events (participants affected / at risk) | 0/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranibizumab (N=49)
Cerebral infarction (Nervous system disorders) | 1 (1) — As the symptom was mild and onset after more than 2 months from the last injection, the serious adverse event (SAE) was categorized as 'Probably not' and reported to the Institutional Review Board (IRB).
Liver cirrhosis (Gastrointestinal disorders) | 1 (2) — The patient had alcoholic hepatitis, and hospitalized due to worsening of alcoholic liver cirrhosis.

LIMITATIONS AND CAVEATS:
Small number of cases, high rate of follow-up loss. Technical problem with measuring caliber of choroidal new vessels.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No